CLINICAL TRIAL: NCT04310748
Title: Effects of TIVA and Inhalation Anesthesia on Oxidative Stress Factors During Hypotensive Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Nur İncekara, MD, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Zeynep01
Record Dates: First submitted 2020-03-06; First posted 2020-03-17 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Oxidative Stress; Anesthesia
Keywords: Total intravenous anesthesia (TIVA); inhalation anesthesia; Thiol-disulphide; Oxidative stress
MeSH Terms: interventions — Anesthesia, Inhalation

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled prospective study to be performed in 60 patients ASA 1 between the ages of 18-55 who will undergo elective rhinoplasty. History of smoking, alcohol, and drug use, who had a BMI>30 are excluding from the study. BIS and TOF monitoring are performing in all patients undergoing standard anesthesia induction. Patients divided into two groups with closed envelope method; TIVA(Group1) and inhalation anesthesia(Group2). In both, MAP target is determining to be in the range of 50-65 mmHg. Blood sample is collecting and storing to measure TAS, TOS, Catalase, Myeloperoxidase, Total Thiol, Native Thiol and Disulfide parameters, before induction and 5, 30, 60 and 120 minutes after induction. The extubation time is recording. The surgical field opinion and satisfaction assessment and the survey presented to the surgeon, respectively. The patients by following up in the recovery unit for 30 minutes; numerical pain scores and nausea-vomiting scores is recording.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Intravenous Anesthesia(TIVA) (Active Comparator): Anesthesia is maintaining with TIVA (Group 1)
  Interventions: Drug: Total Intravenous Anesthesia(TIVA)
- Inhalation Anesthesia (Active Comparator): Anesthesia is maintaining with inhalation anesthesia (Group 2)
  Interventions: Drug: Inhalation Anesthesia

INTERVENTIONS:
Drug: Total Intravenous Anesthesia(TIVA) — Ventilation of the patients was provided with a mixture of 40% oxygen and 60% air. Along with induction, propofol at a dose of 6-10 mg/kg/hour and remifentanil infusion at a dose of 0.3-0.4 mcg/kg/min were started for the maintenance of anesthesia. Drug concentrations were adjusted to maintain BIS values between 40-60 in the maintenance of anesthesia.
  The MAP target was determined to be in the range of 50-65 mmHg. Blood was collected and stored to measure TAS, TOS, Catalase, Myeloperoxidase, Total Thiol, Native Thiol and Disulfide parameters before and after induction at 5,30,60 and 120 minutes. Hemodynamic data (HR, SBP, DBP, MAP, SpO2) and BIS values of the patients were recorded at 5-minute intervals. The extubation time was recorded. The surgical field opinion and satisfaction assessment were made by Boezaart Scoring and the survey presented to the surgeon, respectively. The patients were followed up for 30 minutes; numerical pain scores and nausea-vomiting scores were recorded
  Other Names: Group 1
  Arms: Total Intravenous Anesthesia(TIVA)
Drug: Inhalation Anesthesia — Ventilation of the patients was provided with a mixture of 40% oxygen and 60% N2O. As soon as mechanical ventilation started, sevoflurane was opened at a concentration of 2-3% with a MAK value of 1.1-1.3. Drug concentrations were adjusted to maintain BIS values between 40-60 in the maintenance of anesthesia.
  The MAP target was determined to be in the range of 50-65 mmHg. Blood was collected and stored to measure TAS, TOS, Catalase, Myeloperoxidase, Total Thiol, Native Thiol and Disulfide parameters before and after induction at 5,30,60 and 120 minutes. Hemodynamic data (HR, SBP, DBP, MAP, SpO2) and BIS values of the patients were recorded at 5-minute intervals. The extubation time was recorded. At the end of the surgery, the surgical field opinion and satisfaction assessment were made by Boezaart Scoring and the survey presented to the surgeon, respectively. The patients were followed up for 30 minutes; numerical pain scores and nausea-vomiting scores were recorded.
  Other Names: Group 2
  Arms: Inhalation Anesthesia

SUMMARY:
Total intravenous anesthesia (TIVA) and inhalation anesthesia are two anesthesia methods that can be preferred for the maintenance of anesthesia. Sevoflurane and propofol are drugs used frequently in these methods. This study aims to investigate and compare the effects of inhalation anesthesia using sevoflurane and TIVA using propofol on oxidative stress in patients undergoing controlled hypotensive anesthesia.

DETAILED DESCRIPTION:
Controlled hypotension is defined as keeping systolic blood pressure in the range of 80-90 mmHg or mean arterial pressure in the range of 50-65 mmHg. Pharmacological and non-pharmacological methods can be used to achieve controlled hypotension. Intravenous anesthetics, inhalation anesthetics, opioids, calcium channel blockers, beta blockers, nitrate derivatives are frequently used drugs for this purpose.

General anesthesia maintenance is applied in two ways: total intravenous anesthesia (TIVA) and inhalation anesthesia. The pharmacokinetic and pharmacodynamic properties of drugs used in both methods are quite different.

Products of the body's oxidant antioxidant balance can be measured by biochemical methods and information about this balance can be obtained. Thiols are the regions of proteins most susceptible to oxidation, and the conversion of thiols to disulfides and oxyacids is the earliest marker of radical-mediated protein oxidation.

Total antioxidant status (TAS) shows the total effect of all antioxidants in the human body and total oxidant status (TOS) shows the total effect of oxidants.

In this study, it was aimed to investigate and compare the effects of inhalation anesthesia using sevoflurane and total intravenous anesthesia using propofol on oxidative stress in rhinoplasty cases under controlled hypotension. This assessment was planned using TAS (total antioxidant status), TOS (total oxidant status), Catalase, Myeloperoxidase (MPO), Total Thiol, Native Thiol and Disulfide parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-55
* Who will undergo elective rhinoplasty
* ASA Physical Status Classification System 1

Exclusion Criteria:

* Patients with a history of smoking,
* Patients with a history alcohol use
* Patients with a history drug use,
* Body Mass Index (BMI)>30
* Patients with allergies to drugs to be used
* Patients who refused to participate in the study Termination Criteria
* Whose blood pressure values are out of the targets determined in 3 consecutive measurements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
TAS (TOTAL ANTIOXIDANE STATUS) | Change from Baseline TAS levels at 2 hours
  Evaluation of the effect of anesthesia technique on oxidative stress by TAS values Plasma TAS levels are measured by a commercial mass developed by Erel. Plasma TAS values are expressed in millimeters with the Trolox value per liter.
  3 ml of blood was taken from the venous cannula inserted before the induction of anesthesia into MiniCollect® tubes. At 5, 30, 60 and 120 minutes after induction, 3 ml of blood was taken from the drug-free arm.The collected blood was centrifuged at 2000 x g for 10 minutes and the separated serum was stored at -80 ° C until the study was performed.
TOS (TOTAL OXIDANE STATUS) | Change from Baseline TOS levels at 2 hours
  Evaluation of the effect of anesthesia technique on oxidative stress by TOS values Measurement for TOS is calibrated with hydrogen peroxide and the results are expressed in micromolar by the hydrogen peroxide value per liter (mmol H2O2 equiv / L).
  3 ml of blood was taken from the venous cannula inserted before the induction of anesthesia into MiniCollect® tubes. At 5, 30, 60 and 120 minutes after induction, 3 ml of blood was taken from the drug-free arm.The collected blood was centrifuged at 2000 x g for 10 minutes and the separated serum was stored at -80 ° C until the study was performed.
Catalase | Change from Baseline Catalase levels at 2 hours
  Evaluation of the effect of anesthesia technique on oxidative stress by catalase values The catalase enzyme converts H2O2 into water and oxygen. Catalase enzyme activity decreases in the amount of H2O2 as a result of the dismutase reaction shown by the enzyme in an environment containing H2O2. Catalase enzyme activity is determined by measuring the change in H2O2 concentration at 240 nm. Unit: Unite / L.
  3 ml of blood was taken from the venous cannula inserted before the induction of anesthesia into MiniCollect® tubes. At 5, 30, 60 and 120 minutes after induction, 3 ml of blood was taken from the drug-free arm.The collected blood was centrifuged at 2000 x g for 10 minutes and the separated serum was stored at -80 ° C until the study was performed.
Myeloperoxidase | Change from Baseline Myeloperoxidase levels at 2 hours
  Evaluation of the effect of anesthesia technique on oxidative stress by Myeloperoxidase values Myeloperoxidase activity is determined by measuring the orange color of o-Dianisidine molecule in oxidized environment with H2O2 at 444 nm colorimetrically. The result is calculated using the molar absorption coefficient of the oxidized o-Dianisidine molecule and defined as Unite / L.
  3 ml of blood was taken from the venous cannula inserted before the induction of anesthesia into MiniCollect® tubes. At 5, 30, 60 and 120 minutes after induction, 3 ml of blood was taken from the drug-free arm.The collected blood was centrifuged at 2000 x g for 10 minutes and the separated serum was stored at -80 ° C until the study was performed.
Parameters of Thiol- Disulphide Homeostasis | Change from Baseline Thiol- Disulphide levels at 2 hours
  Evaluation of the effect of anesthesia technique on oxidative stress by Thiol - Disulphide Homeostasis values Extra reduction of DTNB and further reduction of the disulfide bond produced after the DTNB reaction are prevented. The total thiol content of the sample is measured at 410 nm using the modified Ellman reagent. Native thiol content is subtracted from the total thiol content and half of the difference obtained gives the amount of disulfide bond. Unit: μmol / L.
  3 ml of blood was taken from the venous cannula inserted before the induction of anesthesia into MiniCollect® tubes. At 5, 30, 60 and 120 minutes after induction, 3 ml of blood was taken from the drug-free arm.The collected blood was centrifuged at 2000 x g for 10 minutes and the separated serum was stored at -80 ° C until the study was performed.

SECONDARY OUTCOMES:
Surgical Satisfaction: score | postoperative 1 minute
  At the end of the surgery surgeons evaluated surgical satisfaction. the investigators used surgeon satisfaction score which one is performing like that 1- bad 2-moderate 3-good 4-excellent
Bleeding Scores | postoperative 1 minute
  At the end of the surgery surgeons evaluated bleeding scores. the investigators used bleeding score which one is performing like that 0-No bleeding 1-minor bleeding no aspiration required 2- Minor bleeding, aspiration required 3- minor bleeding, frequent aspiration required, 4-Moderate bleeding, visible only with aspiration 5- Severe bleeding,

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Karaaslan, MD, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Fatih, Istanbul, Turkey (Türkiye)